CLINICAL TRIAL: NCT02186002
Title: Single-center, Double-blind, Placebo-controlled, Randomized, Single-ascending Dose, With Nested Cross-over for Food Effect, to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ACT-451840 in Healthy Subjects (Part A)
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ACT-451840 in Healthy Subjects (Part A)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AC-071-101
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: ACT-451840; Safety; Tolerability; Pharmacokinetics
MeSH Terms: interventions — ACT-451840

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): A single oral dose of 10 mg ACT-451840 or placebo to be administered to subjects in the fasted state. Six subjects are to receive ACT-451840 and 2 subjects to receive matching placebo.
  Interventions: Drug: ACT-451840 10 mg; Drug: Placebo
- Group 2 (Experimental): A single oral dose of 50 mg ACT-451840 or placebo to be administered to subjects in the fasted state. Six subjects are to receive ACT-451840 and 2 subjects to receive matching placebo. If indicated by the pharmacokinetic data obtained in the preceding groups and if not previously performed, a food effect investigation will be conducted after a washout period of at least 7 days. A dose of 50 mg ACT-451840 or placebo is to be administered to subjects in the fed state, followed by the second observation period of 4 days. Six subjects who received ACT-451810 in the fasted state are to receive ACT-451840 in the fed state and 2 subjects who received placebo in the fasted state to receive matching placebo in the fed state.
  Interventions: Drug: ACT-451840 50 mg; Drug: Placebo
- Group 3 (Experimental): A single oral dose of 200 mg ACT-451840 or placebo to be administered to subjects in the fasted state. Six subjects are to receive ACT-451840 and 2 subjects to receive matching placebo. If indicated by the pharmacokinetic data obtained in the preceding groups and if not previously performed, a food effect investigation will be conducted after a washout period of at least 7 days. A dose of 200 mg ACT-451840 or placebo is to be administered to subjects in the fed state, followed by the second observation period of 4 days. Six subjects who received ACT-451810 in the fasted state are to receive ACT-451840 in the fed state and 2 subjects who received placebo in the fasted state to receive matching placebo in the fed state.
  Interventions: Drug: ACT-451840 200 mg; Drug: Placebo
- Group 4 (Experimental): A single dose of 500 mg ACT-451840 or placebo to be administered to subjects in the fasted state, followed by an observation period of 4 days. If indicated by the pharmacokinetic data obtained in the preceding groups and if not previously performed, a food effect investigation will be conducted after a washout period of at least 7 days. A dose of 500 mg ACT-451840 or placebo is to be administered to subjects in the fed state, followed by the second observation period of 4 days. Six subjects who received ACT-451810 in the fasted state are to receive ACT-451840 in the fed state and 2 subjects who received placebo in the fasted state to receive matching placebo in the fed state.
  Interventions: Drug: ACT-451840 500 mg; Drug: Placebo
- Group 5 (Experimental): A single oral dose of 1000 mg ACT-451840 or placebo to be administered to subjects in the fasted state. Six subjects are to receive ACT-451840 and 2 subjects to receive matching placebo. If indicated by the pharmacokinetic data obtained in the preceding groups and if not previously performed, a food effect investigation will be conducted after a washout period of at least 7 days. A dose of 1000 mg ACT-451840 or placebo is to be administered to subjects in the fed state, followed by the second observation period of 4 days. Six subjects who received ACT-451810 in the fasted state are to receive ACT-451840 in the fed state and 2 subjects who received placebo in the fasted state to receive matching placebo in the fed state.
  Interventions: Drug: ACT-451840 1000 mg; Drug: Placebo
- Group 6 (Experimental): A single oral dose of ACT-451840 or placebo to be administered to subjects in the fed state. Six subjects are to receive ACT-451840 and 2 subjects to receive matching placebo. The dose of ACT-451840 to be determined on the basis of the pharmacokinetic results for the previous groups
  Interventions: Drug: ACT-451840 (Dose to be determined); Drug: Placebo

INTERVENTIONS:
Drug: ACT-451840 10 mg — ACT-451840 was provided as dry powder, which was reconstituted as a suspension with 25 mL of tap water
  Arms: Group 1
Drug: ACT-451840 50 mg — ACT-451840 was provided as dry powder, which was reconstituted as a suspension with 25 mL of tap water
  Arms: Group 2
Drug: ACT-451840 200 mg — ACT-451840 was provided as dry powder, which was reconstituted as a suspension with 25 mL of tap water
  Arms: Group 3
Drug: ACT-451840 500 mg — ACT-451840 was provided as dry powder, which was reconstituted as a suspension with 25 mL of tap water
  Arms: Group 4
Drug: ACT-451840 1000 mg — ACT-451840 was provided as dry powder, which was reconstituted as a suspension with 25 mL of tap water
  Arms: Group 5
Drug: ACT-451840 (Dose to be determined) — ACT-451840 was provided as dry powder, which was reconstituted as a suspension with 25 mL of tap water
  Arms: Group 6
Drug: Placebo

SUMMARY:
The primary objective of the study was to evaluate the safety and tolerability of ACT-451840 in healthy male subjects.Secondary objectives were : to investigate the pharmacokinetics (PK) of ACT-451840; to investigate the effect of food on the PK of ACT-451840; to evaluate the urinary excretion of ACT-451840 and to investigate the antimalarial activity of ACT-451840.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure.
* Body mass index (BMI) of 18.0 to 28.0 kg/m2 (inclusive) at screening.
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 45-90 beats per minute (inclusive), measured on the dominant arm, after 5 min in the supine position at screening.
* 12-lead electrocardiogram without clinically relevant abnormalities, measured after 5 min in the supine position at screening.
* Hematology, coagulation, clinical chemistry, and urinalysis test results not deviating from the normal range to a clinically relevant extent at screening.
* No clinically significant findings on the physical examination at screening.
* Negative results from urine drug screen at screening.
* Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.
* Subject covered by Health Insurance system and/or in compliance with the recommendations of the National Law in force relating to biomedical research.
* If the subject's partner could become pregnant, reliable methods of contraception must be used from the time of the first administration of study medication until 3 months following administration of the last dose of study medication.

Exclusion Criteria:

* Known allergic reactions or hypersensitivity to any excipient of the drug formulation(s).
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study drug.
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Documented history of chronic liver or gall bladder disease.
* Documented history of hemolytic anemia.
* Veins unsuitable for intravenous puncture on either arm (e.g., veins that are difficult to locate, access, or puncture, veins with a tendency to rupture during or after puncture).
* Previous exposure to the study medication.
* Treatment with another investigational drug within 3 months prior to screening or participation in more than four investigational drug studies within the 12 months prior to screening.
* Subject in the exclusion period of a previous clinical study.
* Subject who had received more than 4,500 Euros as indemnities for his participation in a biomedical research within the 12 last months, including the indemnities for the present study.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* Excessive caffeine consumption, defined as 800 mg or more per day at screening.
* Smoking within 3 months prior to screening and inability to refrain from smoking during the course of the study.
* Previous treatment with any prescribed or over-the-counter medications (including herbal medicines such as St. John's Wort) within 2 weeks prior to first study drug administration.
* Loss of 250 mL or more of blood within 3 months prior to screening.
* Positive results from the hepatitis (hepatitis B and C) serology, except for vaccinated subjects.
* Positive results from human immunodeficiency virus serology at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure from baseline up to end of study | 4 days
  Blood pressure (systolic and diastolic) and pulse rate will be measured using an automatic oscillometric device, always on the dominant/same arm (i.e., dominant arm right = writing with right hand). Measurements should be recorded from the subject in the supine position after having rested for a 5-minute period.
Change in diastolic blood pressure from baseline up to end of study | 4 days
  Blood pressure (systolic and diastolic) and pulse rate will be measured using an automatic oscillometric device, always on the dominant/same arm (i.e., dominant arm right = writing with right hand). Measurements should be recorded from the subject in the supine position after having rested for a 5-minute period.
Change in pulse rate from baseline up to end of study | 4 days
  Blood pressure (systolic and diastolic) and pulse rate will be measured using an automatic oscillometric device, always on the dominant/same arm (i.e., dominant arm right = writing with right hand). Measurements should be recorded from the subject in the supine position after having rested for a 5-minute period.
Change in body weight from baseline up to end of study | 4 days
  Body weight will be measured using the same weighing scale for all subjects and throughout the study. The weighing scale should have a precision of at least 0.5 kg.
Change in heart rate from baseline up to end of study | 4 days
  Heart rate will be measured using a standard 12-lead electrocardiogram recorded at rest with the subject in the supine position for a 5-minute period. Electrocardiograms will be performed immediately prior to dosing and at 1, 2, 4, 6, 8, 12, 24, 48, and 96 hours post dosing.
Change in PQ/PR interval from baseline up to end of study | 4 days
  PQ/PR interval (time interval from the beginning of the P wave to the beginning of the QRS complex) will be measured using a standard 12-lead electrocardiogram recorded at rest with the subject in the supine position for a 5-minute period. Electrocardiograms will be performed immediately prior to dosing and at 1, 2, 4, 6, 8, 12, 24, 48, and 96 hours post dosing.
Change in QRS interval from baseline up to end of study | 4 days
  QRS interval (time interval from the beginning of the Q wave to the end of the S wave) will be measured using a standard 12-lead electrocardiogram recorded at rest with the subject in the supine position for a 5-minute period. Electrocardiograms will be performed immediately prior to dosing and at 1, 2, 4, 6, 8, 12, 24, 48, and 96 hours post dosing.
Change in QTc interval (time interval from beginning of the Q wave until end of the T wave) according to Fridericia's correction (QTcF interval) from baseline up to end of study | 4 days
  QTcF interval will be measured using a standard 12-lead electrocardiogram recorded at rest with the subject in the supine position for a 5-minute period. Electrocardiograms will be performed immediately prior to dosing and at 1, 2, 4, 6, 8, 12, 24, 48, and 96 hours post dosing. The QTcF interval is the QTc interval corrected for heart rate with Fridericia's formula (QTcB = QT/RR^0.33 where RR is 60/heart rate)
Change in QTc interval (time interval from beginning of the Q wave until end of the T wave) according to Bazett's correction (QTcB interval) from baseline up to end of study | 4 days
  QTcB interval will be measured using a standard 12-lead electrocardiogram recorded at rest with the subject in the supine position for a 5-minute period. Electrocardiograms will be performed immediately prior to dosing and at 1, 2, 4, 6, 8, 12, 24, 48, and 96 hours post dosing. The QTcB interval is the QTc interval corrected for heart rate with Bazett's formula (QTcB = QT/RR^0.5 where RR is 60/heart rate).
Number of treatment-emergent electrocardiogram abnormalities from baseline up to end of study | 4 days
  Treatment-emergent electrocardiogram abnormalities will be identified using a standard 12-lead electrocardiogram recorded at rest with the subject in the supine position for a 5-minute period. Electrocardiograms will be performed immediately prior to dosing and at 1, 2, 4, 6, 8, 12, 24, 48, and 96 hours post dosing.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-451840 | 4 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-451840 and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, and 96 hours after dosing.
  Cmax will be calculated on the basis of the blood sampling time points.
Time to maximum plasma concentration (tmax) of ACT-451840 | 4 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-451840 and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, and 96 hours after dosing.
  tmax will be calculated on the basis of the blood sampling time points.
Area under the plasma concentration-time curve (AUC(0-t)) of ACT-451840 | 4 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-451840 and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, and 96 hours after dosing.
  AUC(0-t) will be calculated as the area under the plasma concentration-time profile from time zero to time t of the last measured concentration above the limit of quantification.
Area under the plasma concentration-time curve (AUC(0-infinity)) of ACT-451840 | 4 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-451840 and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, and 96 hours after dosing.
  AUC(0-infinity) will be calculated by combining AUC(0-t) and AUC(extra). AUC(extra) represents an extrapolated value obtained by Ct/λz, where Ct is the last plasma concentration measured above the limit of quantification and λz represents the terminal elimination rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal elimination phase.
Plasma half life (t1/2) of ACT-451840 | 4 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-451840 and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, and 96 hours after dosing.
  t1/2 will be calculated on the basis of the blood sampling time points.
Dose proportionality of single doses of ACT-451840 | 4 days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ACT-451840 and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, and 96 hours after dosing.
  Dose proportionality will be explored by the power model as described by Gough et al [1995]. The power model will be applied to the loge AUC0-∞ and Cmax data. A point estimate and 90% Confidence Interval (CI) will be produced for the population mean slope. Approximate dose proportionality will be concluded if the 90% CI for the slope is completely contained in the range (1+log(0.5))/log(r), 1+log(2)/log(r) where r = high dose/low dose.
Percentage of administered ACT-451840 excreted unchanged in urine | 4 days
  A baseline urine sample will be collected from each subject in the selected dose group after admission on Day -1. On Day 1, subjects will be instructed to empty their bladder immediately prior to study drug intake. Thereafter, all urine produced will be collected during the 4 days following study drug intake until the morning of Day 5. On Day 1, urine will be collected at three consecutive 8-hour intervals, from 0-8 hours, 8-16 hours, and 16-24 hours. On Days 2, 3, and 4 urine will be collected in 24-hours intervals.
Anti-malarial half-maximal inhibitory concentration (IC50) of ACT-451840 | 4 days
  Blood (2.5 mL) will be collected by direct venipuncture or via an intravenous catheter placed in an antecubital vein in the arm into 3.5 mL vacutainer serum separation tubes. The anti-malarial IC50 of ACT-451840 will be determined using a bioassay and ACT-451840 IC50 concentrations will be estimated based on the measured antimalarial activity.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- OPTIMED Clinical Research, Gières, France

REFERENCES:
- [Derived] Bruderer S, Hurst N, de Kanter R, Miraval T, Pfeifer T, Donazzolo Y, Dingemanse J. First-in-humans study of the safety, tolerability, and pharmacokinetics of ACT-451840, a new chemical entity with antimalarial activity. Antimicrob Agents Chemother. 2015 Feb;59(2):935-42. doi: 10.1128/AAC.04125-14. Epub 2014 Nov 24. PMID 25421475